CLINICAL TRIAL: NCT06729944
Title: Diagnostic Value of Next-Generation Sequencing Analysis in Biliary Tract Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BILgenetics_2022; RC 2022-2024 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-12-01; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Hepatectomy; NGS; Stenosis of Bile Duct
Keywords: Next Generation Sequencing; Stenosis of bile duct

STUDY DESIGN:
Intervention Model Description: The patients' biological sample will be analysed by NGS and the results obtained will be compared with the morphological data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing biliary tract resection (Experimental): Patients undergoing biliary tract resection, as part of the normal care pathway, will be enrolled
  Interventions: Diagnostic Test: NGS

INTERVENTIONS:
Diagnostic Test: NGS — Tissue samples will be processed and analysed at the U.O. of Pathological Anatomy

SUMMARY:
The aim of this study is to identify a dysplasia- and CCA-specific NGS panel to increase the diagnostic sensitivity of histological and/or cytological examination of biliary tract stenosis.

DETAILED DESCRIPTION:
Patients undergoing biliary tract resection, as part of the normal course of care, at the O.U. General Surgery and Transplantation will be enrolled. Tissue samples will be processed and analysed at the O.U. of Pathological Anatomy.

Clinical, serological and instrumental data from patients, considered necessary for the intended analyses, will be collected for the purposes of the study.

The study will have a total duration of 36 months. It is planned to enrol 50 patients, all belonging to the U.O. Hepatobiliary and Transplant Surgery of the IRCCS Azienda Ospedaliero-Universitaria di Bologna. The size of the population is estimated on the basis of the number of cases/year from the U.O. Hepatobiliary and Transplant Surgery, and is considered sufficient to achieve the primary objective, since it is an exploratory study. Surgical material (resection of biliary tract, possibly hepatectomy or duodenocephalopancreasectomy), which will be sampled according to clinical practice and sent to the O.U. of Pathological Anatomy of the IRCCS AOUBO, where it will be sampled, fixed in formalin, included in paraffin and processed. From paraffin blocks (selected from those obtained from the sampling of surgical pieces according to clinical practice) 2 µm sections will be cut for Next Generation Sequencing investigations.

ELIGIBILITY:
Inclusion Criteria:

* Availability of enough tissue for histological and NGS analysis (at least 20 ng DNA).
* Age greater than/equal to 18 years.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Identification of an NGS panel specific to dysplasia and CCA | During enrollment period, up to 30 months
  Ratio between the number of cases identified with NGS panel and the number of cases identified with standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Vasuri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No